CLINICAL TRIAL: NCT00989521
Title: Double-blind, Placebo-controlled Crossover Evaluation of the Effect of PUR003 on Subjects With Asthma
Brief Title: Effect of PUR003 on Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pulmatrix Inc. (Industry)
Collaborators: St. Joseph's Healthcare Hamilton / Firestone Institute for Respiratory Health (Unknown); McMaster University (Other)
Responsible Party: Parameswaran Nair, MD, PhD, FRCP, FRCPC, Firestone Institute for Respiratory Health
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 601-1V2
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Asthma; Lung Diseases; Bronchial Diseases
Keywords: Asthma; bronchial diseases; lung diseases; bronchitis; respiratory tract diseases
MeSH Terms: conditions — Asthma; Lung Diseases; Bronchial Diseases; Bronchitis; Respiratory Tract Diseases | interventions — PUR003

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): normal saline for inhalation
  Interventions: Drug: Placebo
- PUR003 (Active Comparator): PUR003 for inhalation
  Interventions: Drug: PUR003

INTERVENTIONS:
Drug: PUR003 — PUR003 for inhalation
  Arms: PUR003
Drug: Placebo — Normal saline for inhalation
  Arms: placebo

SUMMARY:
PUR003 is an inhaled substance that is proposed to assist in the treatment of asthma.

Study objectives are to :

1. to evaluate the safety of PUR003 in subjects with asthma, and
2. to evaluate the efficacy of PUR003 in assisting the treatment of asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Ability and willingness to return to the outpatient clinic for repeated clinic visits and complete all assessments.
3. Adult male or female subject, 18-60 years of age.
4. Stable, mild asthma not requiring any medical treatment other than short acting inhaled bronchodilators, as needed.
5. No smoking within six months prior to entry
6. Must be medically stable.
7. Female subjects must have a negative pregnancy test
8. Subjects of child bearing potential should be sexually inactive (abstinent) for 14 days prior to the first dose of study medication or using an acceptable form of birth control methods.

Exclusion Criteria:

1. History or presence of significant co-existing chronic diseases.
2. History of asthma exacerbations or upper or lower respiratory illness (viral respiratory syndrome, bronchitis, pneumonia) within four weeks of first visit.
3. Pregnancy, breastfeeding.
4. Abused alcohol or illicit drugs that required treatment.
5. Participated in any other investigational drug evaluation within last 30 days.
6. Scheduled to have elective or invasive medical intervention, procedure, or surgery within 6 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2009-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of PUR003 as determined by incidence of adverse events (AEs); changes in physical examination, chest examination; pulmonary function; vital signs; electrocardiogram (ECG) and clinical laboratory assessments. | after three doses

CONTACTS AND LOCATIONS:
Overall Officials: Parameswaran Nair, MD, PhD, Principal Investigator — St. Joseph's Healthcare Hamilton / Firestone Institute for Respiratory Health
Locations (1):
- Firestone Institute for Respiratory Health, Hamilton, Ontario, Canada